CLINICAL TRIAL: NCT01175759
Title: Evaluation of the Efficacy and Safety of the EVE- Skin-Test Panel in Detecting Sensitivity to Sex Hormones in Women With Unexplained Recurrent Pregnancy Loss
Brief Title: Role of Hypersensitivity to Female Sex Hormones in Women With Unexplained Recurrent Pregnancy Loss
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EVE Medical Systems Ltd. (Industry)
Collaborators: Semmelweis University (Other)
Responsible Party: Dr. Yonit Bomstein, EVE Medical systems Ltd.
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 34/2009
Record Dates: First submitted 2010-06-15; First posted 2010-08-05 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-06

CONDITIONS: Abortion, Recurrent
Keywords: Unexplained Recurrent Pregnancy Loss; Recurrent Abortions; Recurrent Miscarriages; Hormones; Skin tests; Allergen; Immunotherapy; Hypersensitivity; Skin reaction
MeSH Terms: conditions — Abortion, Habitual; Hypersensitivity

ARMS (2):
- Healthy control group (Experimental)
  Interventions: Drug: Skin test panel
- UPRL (Experimental)
  Interventions: Drug: Skin test panel

INTERVENTIONS:
Drug: Skin test panel — Skin testing 4 sex hormones will be performed during the luteal phase of the subject's menstrual cycle by study investigators.
  Hormones:
  1. Progesterone 1mmol/L
  2. Estradiol 1mmol/L
  3. Estrone 3mmol/L
  4. Estriol 3mmol/l
     Controls:
  5. Saline (NaCl) 0.9%
  6. Ethyl Oleate with 10% Benzyl Alcohol
  7. Histamine phosphate 1mg/ml (epicutaneous- prick test)
  Arms: Healthy control group
Drug: Skin test panel — Skin testing 4 sex hormones will be performed during the luteal phase of the subject's menstrual cycle by study investigators.
  Hormones:
  1. Progesterone 1mmol/L
  2. Estradiol 1mmol/L
  3. Estrone 3mmol/L
  4. Estriol 3mmol/l
     Controls:
  5. Saline (NaCl) 0.9%
  6. Ethyl Oleate with 10% Benzyl Alcohol
  7. Histamine phosphate 1mg/ml (epicutaneous- prick test)
  Arms: UPRL

SUMMARY:
The EVE- technology is intended for determination of intolerance or sensitivity to female sex hormones among women with hormone-related conditions and for further treatment by desensitization procedure inducing a tolerance to the hormones the women are sensitive to.

This study is designed to evaluate the safety and the ability of the EVE- Skin-Test Panel to detect sensitivity to female sex hormones in subjects with Unexplained Recurrent Pregnancy Loss (URPL) and in Control parous, healthy women.

The Skin Test Panel includes four female hormones and three control solutions.

Hormones from the Skin Test Panel are injected intradermally during the luteal phase of the subject's menstrual cycle. The skin reactions are examined by physician for erythema and wheal after 20 minutes and 48 hours and self-assessed by the patient daily for the following month.

Skin response monthly data is analyzed and compared between unexplained recurrent pregnancy loss (UPRL) and healthy groups.

Following achievement of the significant differences between both groups the immune profile of the healthy and UPRL subjects will be investigated.

ELIGIBILITY:
Inclusion Criteria:

For both groups:

1. Between ages of 20 to 40
2. Willing to participate as shown by signing the informed consent form.

For healthy group:

Parous subjects without premenstrual syndrome, as per medical history and subject's report ( PMS questionnaire)

For UPRL:

Women with three or more documented early pregnancy losses.

Exclusion Criteria:

For both groups:

1. No hormonal contraceptives (either OC or hormonal IUD (Mirena)), no psychotropic agents (e.g. Antidepressants, anxiolytics, or lithium carbonate) for at least two months prior to screening.
2. No hormonal therapy (estrogen or progesterone) for at least two months prior to screening.
3. Significant medical or psychiatric disease.
4. Severe allergies or an inflammatory illness at the time of enrollment

For healthy group:

1. Women who are pregnant or lactating on the day of screening
2. Abnormal routine blood tests

For UPRL:

1. Hereditary thrombophilias (Factor V Leiden, Activated protein C resistance, MTHFR (C677T), Factor II mutation (G20201A))
2. One or more abnormal test from the list below:

   1. Karyotype of either parent (normal: 46XX or 46XY)
   2. Glucose tolerance test (This can be altered to fasting blood sugar of 100mg/dl or less);
   3. Toxoplasmosis serology (IgM positive);
   4. Hysterosalpingogram, 3-D ultrasound or hysteroscopy, thereby excluding anatomical abnormalities, intrauterine adhesions and cervical incompetence;
   5. Thyroid function (Euthyroid levels;);
   6. Serum prolactin;
   7. Normal luteal phase of at least 12 days and plasma progesterone above 24 ng/lL
   8. Anti nuclear factor (Negative)
   9. Anticardiolipin antibody by Elisa testing (cut off value <13 GPLu/mL and <7.6 MPLu/mlL) and Lupus anticoagulant (according to Kaolin clotting time (KCT), Russell's viper venom tome (RVVT) or APTT.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with positive wheal responses to the Skin Test Panel in URPL and Control groups | 1 month

SECONDARY OUTCOMES:
Frequency and severity of adverse events following a skin test procedure in subjects from URPL and Control groups | 1 month
Measurement of cytokine production in subjects from UPRL and Control groups | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: János Rigó, Prof., Principal Investigator — Gynecology and Obstetrics Dept, Semmelweis University, Budapest, Hungary; Henriette Farkas, Prof., Principal Investigator — 3rd Dept of Internal Medicine, Semmelweis University, Budapest, Hungary
Locations (1):
- Depts. Gynecology and Obstetrics and 3rd Dept of Internal Medicine, Budapest, Hungary